CLINICAL TRIAL: NCT06928285
Title: Community Rollout of Technology Enriched Rehabilitation After Stroke: An Implementation Study
Acronym: CROFTERS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Strathclyde (Other)
Collaborators: NHS Lothian (Other Government); NHS Lanarkshire (Other Government); Dundee Leisure and Culture (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UoS_CROFTERS_Kerr2025
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: rehabilitation; technology; implementation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Implementation study assessing;
  1. ability to sustainably deliver NICE (National Institute for Clinical Effectiveness, UK) recommendations for rehabilitation after stroke (intensity and dose)
  2. Response from participants including changes to mobility, communication and impact on life. This will include a data linkage control group with dat aopn health and care use
Masking Description: No masking is used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Technology enriched rehabilitation: Intervention (Experimental): People well enough to exercise lightly but living with motor impairment following a stroke will attend a personalised circuit based programme in a technology enriched rehabilitation gym with exercise and activities structured around their motor, communication and cognitive impairments.
  Interventions: Other: Technology Enriched Rehabilitation

INTERVENTIONS:
Other: Technology Enriched Rehabilitation — The intervention is an 8-week long rehabilitation programme delivered entirely through technology, including virtual reality (immersed and non-immersed), treadmills, weight suspension and movement resistance, and power assistance equipment located in a gym-like space on a university campus. Individual programs are designed, supervised, and reviewed by a physiotherapist using principles of intensity, feedback, cognitive engagement, and aerobic activity to address the goals identified by the participant and scores from outcome measures at baseline. Participants should attend a minimum of two times per week and can more frequently for the two hour group based circuit class.

SUMMARY:
The minimum guideline recommendations for rehabilitation after stroke are not being met. This compromises individual recovery and increasing the global burden of disability. A multi-technology solution, co-created with people living with stroke, has been shown to be feasible in both sub-acute and chronic populations but has not been implemented as an integrated rehabilitation service.

The aim of this implementation study is to assess the ability of a technology enriched model of rehabilitation to deliver guideline recommendations in a range of NHS and local authority settings that provide rehabilitation services to stroke survivors at different stages of their recovery. The findings will be used to co-create a scalable, adaptable, and sustainable model that meets rehabilitation guidelines.

DETAILED DESCRIPTION:
A recently completed pilot study (NCT05981729) demonstrated the feasibility of our multi-technology circuit based model of rehabilitation in an acute NHS stroke unit (UHW, NHS Lanarkshire). The key findings were that the model delivered an average of 52 minutes of additional rehabilitation every day, without any safety concerns and with supervision provided by rehabilitation assistants. Importantly for future implementation the participating patients and ward staff were all very positive about the novel approach. The challenge now is to translate these positive findings into a sustainable national solution that maintains fidelity to the key parameters of evidence-based rehabilitation (personalised, high intensity, and enriched environment) and can be adopted by diverse service providers (NHS, Local Authority, and medical charities) across various settings, to support people through their whole recovery journey.

Aim To develop an acceptable and sustainable implementation model of technology enriched rehabilitation after stroke that sustainably delivers NICE (National Institute for Clinical Effectiveness) guideline recommendations in a range of rehabilitation settings and phases of recovery after stroke.

Design This is an implementation study using a mixed methods approach to assess technology enriched rehabilitation gyms across a network of NHS, local authority and 3rd sector funded rehabilitation services. Part of the implementation study will involve gathering preliminary evidence of efficacy through comparison with a control group matched for age and stroke through a data linkage project (eDRIS, Data Scotland).

Locations Four locations have agreed to participate, they represent different stages of recovery after stroke, from acute illness (University Hospital Wishaw, Wishaw, UK) to community care (Blantyre Life, Blantyre, UK) and Edinburgh Community Stroke Service, Edinburgh, UK) and long-term maintenance (Olympia leisure centre, Dundee, UK). At one location (Edinburgh) the study will also test whether a higher dose of rehabilitation can be delivered within current resources including participant tolerance and what resources are required to maintain a high dose delivery.

Participants All participants will have a diagnosis of stroke (physician diagnosed) and be suitable for rehabilitation. Specific eligibility criteria, such as time since stroke, will vary across the locations and are detailed later.

Intervention This will be delivered by the local teams of suitably qualified (e.g. physiotherapists) staff following training from the Strathclyde team.

Intervention parameters Frequency: at least twice a week Intensity: Always sub-maximal. Determined by the amount of time spent in each activity and (where possible) the number of movements (e.g. steps on treadmill) performed Time: 2 hours max with activities varied between seated and standing Total duration: 8 weeks

Content

The TERG intervention has been described in general terms in recent publications (Kerr, Grealy et al. 2021, Kerr, Keogh et al. 2023) and is detailed in a comprehensive manual which will be used for training and to improve fidelity. The key elements are described below:

Once consent has been taken and outcome measures have been recorded each participant should be supported in setting three personal goals. Some training will be provided around effective goal setting. These, together with the initial outcome measures, will be used to structure an initial training programme that will be reviewed regularly (every 2 weeks). The programme will only use the technology listed below and individuals should be trained (as much as possible) to use the equipment on their own, with physical assistance and support provided by the supervising staff.

Rehabilitation equipment and purpose:

1. Treadmill with adjustable walking harness system. Purpose: Gait and balance training
2. Large, height adjustable, computer tablet with digital health apps. Purpose: Communication and cognitive training performed in standing or sitting
3. GripAble hand trainer. Purpose: Upper limb training and cognitive training
4. Mirror Therapy. Purpose: Motor priming & upper limb training
5. Power assisted Seated rower. Purpose: General exercise, aerobic, strength, flexibility
6. Power assisted Cross cycle trainer. Purpose: General exercise, aerobic, strength, flexibility
7. Power assisted Seated climber. Purpose: General exercise, aerobic, strength, flexibility
8. Power assisted bike: Purpose: General exercise, aerobic, strength, flexibility
9. VR headset; Purpose: Upper limb and balance upper limb co-ordination and balance

On completion of the 8 week programme outcome measures will be repeated and participants will be interviewed by a researcher not involved in the programme delivery to understand the user experience.

Data collected

1. Participant attendance (number sessions attended) and engagement (movements performed) with activities.
2. Incidence of safety events (adverse events)
3. Interviews with staff and participants
4. Delivery costs (staff and equipment)
5. Standard measures of mobility (10 mwt, five times sit to stand), communication and patient reported outcomes on function (Rivermead Mobility Index) and quality of life (Stroke Impact Scale). These will be recorded before the programme begins and immediately after completion.
6. Health and Care costs for 6 months after intervention through a data linkage project

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* Currently well
* Suitable for rehabilitation (motor/ciommunication and or/cognitive impairment(
* Able to attend the programme for two hours at least twice a week
* Able to follow instructions in English and follow provide verbal and/or written feedback

Exclusion Criteria:

* Absolute contradictions to physical activity
* Recent (6 weeks) deterioration in health
* Change in medication
* Currently unwell

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
10-meter walk test (10mWT) | Three time points; 1) Two weeks before intervention starts at the initial induction meeting,2) immediately before the intervention, and 4) immediately after intervention ends
  Time to walk 10 metres
Five times sit to stand movement | Three time points; 1) Two weeks before intervention starts, at the induction meeting,2) immediately before the intervention and 3) immediately after intervention ends
  Time to complete five sit to stand movements safely.

SECONDARY OUTCOMES:
Stroke Impact Scale | Two time points; 1) Two weeks before intervention starts and 2) immediately after intervention ends
  Quality of life index for people after stroke
Action Research Arm Test (ARAT) | Two time points; 1) Two weeks before intervention starts and 2) immediately after intervention ends
  19 item observational measure to assess upper extremity performance (coordination, dexterity and functioning) after stroke

OTHER OUTCOMES:
Communication Outcome after Stroke (COAST) scale | Two time points; 1) Two weeks before intervention starts and 2) immediately after intervention ends
  Patient-centred measure of communication effectiveness for people with aphasia after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Kerr, PhD, Study Director — University of Strathclyde

IPD SHARING:
Plan to Share IPD: Yes
We will share the outcomes of the implementation study including interview transcipts and outcome measures
Supporting Information: Study Protocol, CSR
Time Frame: August 2027 for 5 years
Access Criteria: This will be publicly available from the University of Strathclyde repository (PURE)
URL: https://www.strath.ac.uk/research/researchdatamanagementsharing/datadeposit/